CLINICAL TRIAL: NCT07206836
Title: Comparison of Outcome of Colostomy Reversal in Pediatric Patients With Enhanced Recovery After Surgery Versus Traditional Care Protocols.
Brief Title: Pediatric Colostomy Reversal: Traditional Care vs. Enhanced Recovery After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Salman Ali, Post-Graduate Resident, Children Hospital Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 696/CH&ICH/FSD
Record Dates: First submitted 2025-09-13; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Colostomy - Stoma; Stoma Reversal Procedure; ERAS
Keywords: Pediatric Colostomy; Colostomy Reversal; Enhanced Recovery After Surgery; ERAS; Traditional Care protocol; Length of Hospital Stay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Recovery after Surgery (ERAS) (Experimental): Patients undergoing colostomy reversal managed with the Enhanced Recovery After Surgery (ERAS) protocol, which emphasizes reduced fasting, avoidance of mechanical bowel preparation, early postoperative oral feeding, and multimodal non-opioid analgesia.
  Interventions: Other: Enhanced Recovery after Surgery Protocol
- Traditional Care Protocol (Active Comparator): Patients undergoing colostomy reversal managed with the traditional perioperative care protocol, including three days of mechanical bowel preparation, overnight fasting before surgery, routine nasogastric tube placement, opioid-based postoperative pain control, and delayed resumption of oral intake.
  Interventions: Other: Traditional Care Protocol

INTERVENTIONS:
Other: Enhanced Recovery after Surgery Protocol — reduced fasting, no mechanical bowel prep, early feeding, non-opioid analgesia.
  Other Names: ERAS
  Arms: Enhanced Recovery after Surgery (ERAS)
Other: Traditional Care Protocol — Participants receive standard peri-operative management for colostomy reversal. This includes three days of mechanical bowel preparation with oral laxatives and clear fluids, overnight fasting before surgery, routine nasogastric tube placement, opioid-based postoperative pain control, and a nil-per-mouth regimen for at least three days after surgery before gradually resuming oral intake.
  Arms: Traditional Care Protocol

SUMMARY:
The goal of this clinical trial is to learn whether using an Enhanced Recovery After Surgery (ERAS) protocol helps children recover faster after colostomy reversal compared with traditional care.

The main question it aims to answer is:

Does ERAS lower the number of days children need to stay in the hospital after colostomy reversal compared with traditional care?

Researchers will compare two groups:

ERAS group - Children receive shorter pre-surgery fasting, no mechanical bowel preparation, early pain control, and early feeding after surgery.

Traditional care group - Children receive the usual long bowel preparation, overnight fasting, opioid pain medicine, and a longer period without food after surgery.

Participants will:

Be randomly assigned to either the ERAS or traditional care group

Have their colostomy surgically closed by experienced pediatric surgeons

Be monitored daily until they can eat a solid meal without vomiting; this marks the end of their hospital stay

The study will enroll 60 children ages 2-13 at Children's Hospital Faisalabad, Pakistan.

Researchers will measure length of hospital stay from surgery until discharge as the main outcome.

DETAILED DESCRIPTION:
This single-center, prospective randomized controlled trial will compare two perioperative care strategies for pediatric colostomy reversal: the Enhanced Recovery After Surgery (ERAS) protocol and the conventional Traditional Care Protocol (TCP). The study is being conducted in the Department of Pediatric Surgery at the Children's Hospital and Institute of Child Health, Faisalabad, Pakistan.

Scientific Rationale

Colostomy reversal restores bowel continuity after temporary fecal diversion, which is frequently performed in children with anorectal malformations (ARM), Hirschsprung's disease (HD), or following severe perineal injury. Conventional postoperative care has historically included three days of mechanical bowel preparation, prolonged pre-operative fasting, routine nasogastric decompression, opioid-based analgesia, and delayed oral feeding. Evidence from both adult and pediatric literature shows that ERAS protocols-emphasizing minimal bowel preparation, shortened fasting, multimodal non-opioid analgesia, and early enteral feeding-can reduce hospital stay and enhance recovery without increasing complications. However, high-quality pediatric data, especially from South Asia, remain limited.

Study Design

The trial will enroll 60 children (ages 2-13 years) who meet inclusion criteria and have no major comorbidities or prior extensive abdominal surgery. Using a computer-generated randomization table, participants will be allocated in a 1:1 ratio to either the ERAS or TCP arm. The allocation will occur after informed consent from parents or guardians.

ERAS arm:

Pre-operative preparation consists of two rectal enemas and oral laxative 12 hours apart on the day before surgery.

Clear oral fluids are allowed until three hours prior to anesthesia.

Intraoperative management includes minimal bowel handling and caudal block for pain control.

Postoperative care features avoidance of opioid analgesia, removal of nasogastric tube within 48 hours, and initiation of clear oral fluids followed by early progression to solid diet as tolerated.

Traditional Care arm:

Mechanical bowel preparation and clear fluid diet for three days before surgery.

Overnight fasting and intra-venous antibiotics are given.

Postoperative management includes routine nasogastric decompression with a nil-per-mouth regimen for at least three days, opioid analgesia, and gradual reintroduction of oral intake starting on postoperative day three or four.

All operations will be performed by consultant pediatric surgeons with at least five years of post-FCPS experience to ensure procedural consistency.

Data Collection and Analysis

Daily postoperative assessments will include vital signs, abdominal examination, and tolerance of oral intake. Laboratory evaluation on postoperative day one will include complete blood count and serum electrolytes, with corrections as indicated. The primary endpoint is length of hospital stay, defined as the number of days from surgery to discharge once the child consumes at least one age-appropriate solid meal without vomiting for six hours. Data will be entered in SPSS version 25. Quantitative variables will be summarized as means and standard deviations; qualitative variables as frequencies and percentages. Independent-sample t tests will compare the primary outcome between groups. Age, gender, and underlying diagnosis will be assessed as potential effect modifiers through stratification followed by post-stratification t tests. A p-value ≤0.05 will be considered statistically significant.

Significance

This study addresses a key evidence gap by providing randomized controlled data on ERAS in a high-volume pediatric surgical setting in Punjab, Pakistan. Demonstrating a reduction in hospital stay without added complications could support broader adoption of ERAS protocols, improving patient turnover, reducing healthcare costs, and enhancing recovery for children undergoing colostomy reversal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Colostomy
* Admitted for Reversal of colostomy

Exclusion Criteria:

* Patients with endocrinal abnormalities
* Patients with cardiac abnormalities
* Patients with spinal abnormalities
* Patients with bleeding abnormalities
* Patients who have undergone previous multiple abdominal surgeries

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay (Days) | From date of surgery through hospital discharge (an average of 3-14 days)
  Duration of hospitalization measured from the day of surgery until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital and Institute of Child Health Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Age, Gender, Diagnosis, Arm of study, Length of Hospital Stay
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and supporting documents (study protocol and statistical analysis plan) will be available beginning 6 months after publication of the primary results and for a period of 3 years thereafter
Access Criteria: De-identified data will be shared with qualified researchers who submit a methodologically sound proposal to address a scientifically valid question. Requests should be sent to SalmanAli@live.com. Access will be granted after approval by the principal investigator and ethics committee. Data will be provided through a secure, password-protected platform for research use only and must not be used to re-identify participants.